CLINICAL TRIAL: NCT01883817
Title: Docosahexaenoic Acid Augmentation of Cortical Attention Networks in ADHD
Brief Title: Effect of Omega-3 Fatty Acid on Cortical Function in ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Principal Investigator, Robert McNamara, Associate Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013-0199
Record Dates: First submitted 2013-06-06; First posted 2013-06-21 (Estimated); Results first posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-02

CONDITIONS: Attention Deficit Disorder
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Docosahexaenoic Acids; Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Corn/soy oil placebo capsules that are similar in shape and color to the DHA capsules given over 10 weeks
  Interventions: Drug: Placebo
- DHA Omega-3 (Experimental): Long-chain omega-3 fatty acid docosahexaenoic acid (DHA) at 1,200 mg/day, 600 mg twice daily for 10 weeks
  Interventions: Drug: DHA Omega-3

INTERVENTIONS:
Drug: DHA Omega-3 — Patients will receive a fixed dose of DHA (1,200 mg/day, 600 mg twice daily) or placebo (corn/soy oil) over 10 weeks
  Other Names: Docosahexaenoic acid; Omega 3 Fatty Acids
  Arms: DHA Omega-3
Drug: Placebo — corn/soy oil capsule with similar color, taste, and shape as experimental drug (DHA)
  Other Names: Inactive drug
  Arms: Placebo

SUMMARY:
The study hypothesis is that DHA is more effective than placebo in increasing brain activation and reducing symptoms in psychostimulant-free children with ADHD.

DETAILED DESCRIPTION:
This study aims to determine the effects of 10-week dietary supplementation with the long-chain omega-3 fatty acid docosahexaenoic acid (DHA) or placebo on prefrontal cortical structural and functional connectivity using several neuroimaging techniques: DTI (Diffusion Tensor Imaging), 1H MRS(Proton Magnetic Resonance Spectroscopy), and fMRI (Functional Magnetic Resonance Imaging) in psychostimulant-free children with attention deficit hyperactivity disorder (ADHD). It is postulated that DHA supplements will increase brain activation and reduce ADHD symptomatology.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent/assent
* Ages 5-15 years old
* Meets DSM-IV-TR criteria for ADHD as determined by the KSADS

Exclusion Criteria:

* Contraindication to an MRI scan (i.e., braces, claustrophobia)
* A history of a major medical (e.g., diabetes) or neurological illness (e.g., epilepsy)
* Greater than 1 year outside appropriate age/grade level
* A history of intolerance or hypersensitivity to omega-3 fatty acids
* Currently taking omega-3 supplements
* Not proficient in English language
* Any history of a hematological disorder or concomitant use of anticoagulant medications
* Personal history of an Axis I psychiatric disorder other than ADHD
* Inability to swallow capsules

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2017-03-03 (Actual); Study Completion 2017-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert K McNamara, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Department of Psychiatry and Behavioral Neuroscience, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | DHA Omega-3
Started | 14 | 16
Completed | 10 | 9
Not Completed | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Corn/soy oil placebo capsules that are similar in shape and color to the DHA capsules given over 12 weeks
  Placebo: corn/soy oil capsule with similar color, taste, and shape as experimental drug (DHA)
- DHA Omega-3: Long-chain omega-3 fatty acid docosahexaenoic acid (DHA) at 1,200 mg/day, 600 mg twice daily for 12 weeks
  DHA Omega-3: Patients will receive a fixed dose of DHA (1,200 mg/day, 600 mg twice daily) or placebo (corn/soy oil) over 12 weeks
- Total: Total of all reporting groups
Arm/Group | Placebo | DHA Omega-3 | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 16 | 30
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 11 | 12 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 7 | 9 | 16
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Attention-Deficit Hyperactivity Disorder Symptom Ratings Using the ADHD Rating Scale (ADHD-RS-IV)
Description: Attention-Deficit Hyperactivity Disorder Rating Scale Version IV (ADHD-RS-IV) Min score: 0 Max score: 54 Higher score = more severe ADHD symptoms
Time Frame: 10 weeks
Population: Adolescents with a current Diagnostic and Statistical Manual of Mental Disorders, 4th edition, Text Revision diagnosis of Major Depressive Disorder or Depressive Disorder not otherwise specified, a Childhood Depression Rating Scale-Revised (CDRS-R) Version raw score of >40, and at least one biological parent with bipolar I disorder.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | DHA Omega-3
Number analyzed (Participants) | 14 | 16
score on a scale | 47.1 (8.5) | 46.1 (6.6)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Placebo | DHA Omega-3
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 0/14 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-06-19): https://cdn.clinicaltrials.gov/large-docs/17/NCT01883817/Prot_SAP_000.pdf